CLINICAL TRIAL: NCT00616018
Title: Acetaminophen Adduct Formation in Alcohol Abstaining Subjects Administered Therapeutic Doses of Acetaminophen for Ten Consecutive Days
Brief Title: Acetaminophen Adduct Formation in Non-Drinkers Taking Therapeutic Doses of Acetaminophen for Ten Consecutive Days
Acronym: Non-Drinker
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kennon Heard (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kennon Heard, Medical Toxicology Fellowship Director, Denver Health and Hospital Authority
Organization: Denver Health and Hospital Authority (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: COMIRB #06-1187; COMIRB #06-1187
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Drug Induced Liver Injury
Keywords: acetaminophen; protein adducts; hepatic function; drug safety; non drinkers
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): all subjects receive 4 g/day of acetaminophen for 10 consecutive days in this open-label study
  Interventions: Drug: acetaminophen

INTERVENTIONS:
Drug: acetaminophen — 4 g/day for 10 consecutive days
  Other Names: Tylenol Extra Strength

SUMMARY:
Acetaminophen is commonly used to treat fever or pain. Your body clears acetaminophen by processing it in the liver. During the processing, some of the acetaminophen may bind to proteins in the liver. The protein-acetaminophen product is called an "adduct." After a large acetaminophen overdose, the liver has to process a lot of acetaminophen, so large amounts of adducts are formed. However, we have found that lower levels may be formed even when people take recommended doses. The purpose of this study is to measure the amount of adducts formed when healthy people who do not drink alcohol take normal doses of acetaminophen for 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. age 21 years or older
2. provide written informed consent
3. consume, on average, less than 1 alcoholic beverage daily for the previous 3 months and would be considered non-drinkers

Exclusion Criteria:

1. History of ingesting more than 4 grams of acetaminophen per day for any of the 4 days preceding study enrollment
2. Currently taking isoniazid
3. Consumption of any alcoholic beverage during the run-in period
4. A detectable serum acetaminophen at baseline
5. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 50 IU/L at the start of the run-in period or at baseline
6. Platelet count less than 125,000/cc at baseline
7. Positive pregnancy test at baseline (female participants only)
8. Currently adheres to a fasting type diet as determined by self report
9. Currently has anorexia nervosa as determined by self report
10. Subject appears clinically intoxicated, psychiatrically impaired or unable to give informed consent for any reason
11. Known hypersensitivity to acetaminophen

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kennon Heard, MD, Principal Investigator — Denver Health/Rocky Mountain Poison & Drug Center
Locations (1):
- Denver Health Rocky Mountain Poison and Drug Center, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted from August 2007 through January 2008. Healthy volunteers were recruited through flyers posted in community settings.
Pre-assignment Details: Thirty-five subjects were consented for the study. Of these, eight were excluded (six did not meet inclusion criteria and two refused to participate). The 27 eligible subjects were assigned to the treatment arm to receive 4 grams of acetaminophen per day, for 10 consecutive days.
Groups:
- Acetaminophen: all subjects receive 4 g/day of acetaminophen for 10 consecutive days in this open-label study
Period: Overall Study
Arm/Group | Acetaminophen
Started | 27
Completed | 24
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Acetaminophen
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Serum Level of Acetaminophen-cysteine (APAP-Cys) Protein Adducts
Description: Acetaminophen-cysteine (APAP-Cys) protein adduct concentrations were measured at Day 0, 4, 7, 9, 11 and 14. All units are in nmol/mL serum.
Time Frame: Day 0, 4, 7, 9, 11, and 14.
Population: Analysis is based upon the 24 subjects who completed all study visits.
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | Acetaminophen
Number analyzed (Participants) | 24
nmol/mL
  Day 0 | 0.0 (0.0)
  Day 4 | 0.3 (0.1)
  Day 7 | 0.3 (0.2)
  Day 9 | 0.4 (0.2)
  Day 11 | 0.4 (0.2)
  Day 14 | 0.2 (0.1)

2. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: ALT was measured at Day 0, 4, 7, 9, 11, and 14.
Time Frame: Day 0, 4, 7, 9, 11, and 14.
Population: Analysis is based upon the 24 subjects who completed all study visits.
Measure: Mean (Standard Deviation); unit: IU/L
Groups:
- Acetaminophen: acetaminophen treatment group
Arm/Group | Acetaminophen
Number analyzed (Participants) | 24
IU/L
  Day 0 | 24.0 (8.1)
  Day 4 | 25.9 (10.1)
  Day 7 | 41.3 (27.3)
  Day 9 | 41.3 (27.3)
  Day 11 | 41.8 (24.2)
  Day 14 | 36.1 (18.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of first dose of study medication through followup visits.
Arm/Group | Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 12/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen (N=27)
diarrhoea (Gastrointestinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 5 (6)
fatigue (General disorders) | 2 (2)
headache (Nervous system disorders) | 3 (6)
migraine (Nervous system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
One limitation is that this study did not include a placebo group. The study was limited to healthy volunteers. The ingestion of each dose and use of other medications was self-reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No